CLINICAL TRIAL: NCT03291951
Title: FOcus on Reducing Dose-limiting Toxicities in Colon Cancer With Resistance Exercise Study
Acronym: FORCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Penn State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CN-17-2877
Record Dates: First submitted 2017-09-07; First posted 2017-09-25 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Resistance Training; Colon Cancer; Chemotherapy Effect
MeSH Terms: conditions — Colonic Neoplasms | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial of resistance training intervention in colon cancer patients receiving chemotherapy consists of two arms: an in-person and telephone-based intervention to promote home-based resistance training, and a wait-list, control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance training group (Experimental): Participants randomized to the resistance training (RT) group will receive an in-person and telephone-based intervention to promote home-based resistance training. The exercise intervention will begin by the 3rd adjuvant chemotherapy visit and continue exercise through the completion of post-operative chemotherapy. Participants will work with an exercise professional with expertise working with oncology patients.
  Interventions: Behavioral: Resistance training
- Usual care group (No Intervention): Participants randomized to the usual care (U) group will be instructed to refer to their physician regarding what forms of exercise are safe for them, given their medical history. The U group will be told to continue whatever exercise program they have been undertaking up to enrolling in the study, but not to increase exercise or begin weight-lifting over the period of study participation.

INTERVENTIONS:
Behavioral: Resistance training — The intervention goal is for study participants to exercise with progressively higher weights for resistance training to achieve a 1-kg increase in lean body mass by the end of the intervention. During an in-person visit on the same day as a chemotherapy infusion session, exercise professionals will teach participants a series of exercises to be completed at home twice weekly throughout the intervention. Participants will also receive protein powder, which they will be instructed to consume with meals twice a day. During subsequent infusion sessions, the exercise professional will meet in-person with participants to evaluate their ability to increase weights, and adjust exercises appropriately. In between visits, the exercise professional will check-in with participants by phone.
  Arms: Resistance training group

SUMMARY:
FORCE is a randomized home-based resistance training/strength training (RT) intervention study for Stage II and III colon cancer patients undergoing chemotherapy.

Participants will be 180 newly diagnosed Stage II and III colon cancer patients from Kaiser Permanente of Northern California (KPNC), the Penn State Cancer Institute (PSCI), and the Dana Farber Cancer Institute (DFCI). The intervention will begin within the first weeks of adjuvant chemotherapy and continue exercise through the completion of post-operative chemotherapy. Specifically, the investigators will examine between group differences for RT versus waitlist control for chemotherapy outcomes including dose delays, dose reductions, early stoppage and Grade 3 and 4 toxicities. The investigators will also study changes in muscle mass (MM) and changes in specific inflammatory markers (e.g. CRP, IL-6 and TNF-RII) as potential markers of change in response to RT. To determine effects of change of MM on chemotherapy-specific drug clearance, the investigators will examine the impact body composition changes on the pharmacokinetics (PK) of 5-FU and oxaliplatin, two of the most commonly used drugs for colon cancer.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥18 years
* Newly diagnosed with histologically confirmed stage II-Ill colon cancer
* Completed curative-intent surgical resection
* Currently prescribed one of the following adjuvant chemotherapy regimens: (IV 5-fluorouracil [5-FU] / leucovorin [LV], capecitabine, FOLFOX [5-FU, LV, oxaliplatin], CAPOX [capecitabine and oxaliplatin]
* Patients must have started chemotherapy or plan to start with receipt of the first exercise visit by 3rd infusion visit. Patients enrolled at the Dana-Farber Cancer Institute and who are receiving FOLFOX chemotherapy are eligible to enroll in the pharmacokinetics sub-study.
* No planned major surgery anticipated in the intervention period
* Sufficient time to heal from any major surgery to start of intervention, including colostomy reversal (port-a-cath removal excluded)
* Approval by either oncologist or surgeon to participate in trial
* Readiness as determined by the Physical Activity Readiness Questionnaire
* Ability to understand and the willingness to sign a written informed consent document in English
* Willingness to be randomized

Exclusion Criteria:

* Concurrent actively treated other cancer (except non-melanoma skin cancer, in situ cervical cancer or localized prostate cancer treated with surveillance only)
* Patients with untreated hypertension (>180 mm Hg systolic or >100 mm Hg diastolic) appearing in the patient's medical record in the two weeks prior to screening
* Presence of metastatic disease
* Current strength training >2x week for the past 3 or more months
* Patients enrolled in other clinical trials of weight loss, physical activity or dietary interventions are ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Relative dose intensity (RDI) | 3-6 months
  Chemotherapy completion rates will be assessed as relative dose intensity for each agent and then average relative dose intensity (ARDI), which considers all chemotherapy agents in a regimen. We will examine differences in RDI for each chemotherapy agent and the ARDI across all agents between the RT group and the UC group.
Number of moderate and severe chemotherapy-associated toxicities | 3-6 months
  Moderate and severe chemotherapy-associated toxicities will be assessed via a NCI PRO-CTCAE questionnaire, which is a patient-reported outcome measure developed to evaluate symptomatic toxicity in patients on cancer clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Bette J Caan, DrPH, Principal Investigator — Kaiser Permanente; Kathryn H Schmitz, PhD, MPH, Principal Investigator — Penn State Cancer Institute; Jeffrey Meyerhardt, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Kaiser Permanente Division of Research, Oakland, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Penn State Cancer Institute, Hershey, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee S, Ma C, Caan BJ, Binder AM, Brown JC, Pena Perez A, Lee C, Weltzien E, Ross MC, Quesenberry CP, Campbell KL, Cespedes Feliciano EM, Castillo A, Schmitz KH, Meyerhardt JA. Impact of resistance training on inflammatory biomarkers and associations with treatment outcomes in colon cancer. Cancer. 2025 May 1;131(9):e35865. doi: 10.1002/cncr.35865. PMID 40278841
- [Derived] Compton SLE, Yang S, Madere J, Weltzien EK, Caan BJ, Meyerhardt JA, Schmitz KH, Brown JC. Dietary quality and chemotherapy-induced peripheral neuropathy in colon cancer. Cancer. 2025 Jan 1;131(1):e35599. doi: 10.1002/cncr.35599. Epub 2024 Oct 5. PMID 39369275
- [Derived] Brown JC, Yang S, Compton SLE, Campbell KL, Cespedes Feliciano EM, Quinney S, Sternfeld B, Caan BJ, Meyerhardt JA, Schmitz KH. Effect of resistance training on physical function during chemotherapy in colon cancer. JNCI Cancer Spectr. 2024 Jul 1;8(4):pkae058. doi: 10.1093/jncics/pkae058. PMID 39012500

DOCUMENTS (3):
  • Study Protocol (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/51/NCT03291951/Prot_001.pdf
  • Statistical Analysis Plan (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/51/NCT03291951/SAP_002.pdf
  • Informed Consent Form (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/51/NCT03291951/ICF_003.pdf